CLINICAL TRIAL: NCT00206583
Title: A Multicenter, Open-label Uncontrolled Study to Investigate the Efficacy and Safety of a 4-phasic Oral Contraceptive SH T0065 in a 28-day Regimen for 13 Cycles in Healthy Female Subjects
Brief Title: Efficacy and Safety Study of an Oral Contraceptive in Healthy Females
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 90959; 304742 (Other: Company internal)
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EV/DNG (Qlaira, BAY86-5027) (Experimental): Estradiolvalerate (EV)/Dienogest (DNG) Tablet p.o. (oral)
  Interventions: Drug: EV/DNG (Qlaira, BAY86-5027, SH T00658ID)

INTERVENTIONS:
Drug: EV/DNG (Qlaira, BAY86-5027, SH T00658ID) — GA: Estradiolvalerate (EV)/Dienogest (DNG) Tablet p.o. (oral) Tablet, p.o. (oral)

SUMMARY:
The purpose of this study is to determine whether the study drug is safe and effective in the prevention of pregnancies in a large group of volunteers.

DETAILED DESCRIPTION:
This study has previously been posted by Berlex, Inc. Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals Inc.. Bayer HealthCare Pharmaceuticals Inc. is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women between the ages of 18 and 35 years requiring contraception

Exclusion Criteria:

* Pregnancy, lactation, and contraindication of combined oral contraceptive

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 499 (Actual)
Dates: Start 2005-03; Primary Completion 2007-06 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Number of unintended pregnancies after 1 year | Throughout 1 year of treatment

SECONDARY OUTCOMES:
Bleeding pattern and cycle control parameters after 1 year | Throughout 1 year of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (29):
- United States (20):
  - Women and Children's Hospital, Los Angeles, Los Angeles, California
  - Lifespan Research, Palo Alto, California
  - Genesis Center for Clinical Research, San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - Harbor - UCLA Medical Center, Torrance, California
  - Clinical Trial Center of Colorado, Castle Rock, Colorado
  - New Age Medical Research Corp., Miami, Florida
  - Visions Clinical Research, Palm Springs, Florida
  - Insignia Care for Women, P.A., Tampa, Florida
  - Comprehensive Clinical Trials, West Palm Beach, Florida
  - Physicians Research Group, Indianapolis, Indiana
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Women's Clinic of Lincoln, PC, Lincoln, Nebraska
  - Women's Care Source, Morristown, New Jersey
  - OB/GYN Health Center, Medford, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Clinical Research of Philadelphia, LLC, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Health System, Pittsburgh, Pennsylvania
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Seattle Women's: Health, Research, Gynecology, Seattle, Washington
- Canada (9):
  - Total Concept Health Care Inc., Kitchener, Ontario
  - Temple Green Clinic, Waterloo, Ontario
  - Rhodin Recherche Clinique, Drummondville, Quebec
  - Centre d'étude clinique de Montréal Inc., Montreal, Quebec
  - Les Gynecologues Associes, Montreal, Quebec
  - Clinique Recherche en Sante des Femmes Inc., Québec, Quebec
  - Clinique de Gynecologie, Shawinigan, Quebec
  - Diex Recherche Inc., Sherbrooke, Quebec
  - Clinique Médicale des Campus, Ste-Foy, Quebec